CLINICAL TRIAL: NCT03641235
Title: Analysis of the Dynamics of the Lung Microbiota During Acute Exacerbation of COPD Requiring Admission to Intensive Care
Brief Title: Analysis of the Dynamics of the Lung Microbiota During Acute Exacerbation of COPD Requiring Admission to Intensive Care Unit
Acronym: ADMiRE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/17
Record Dates: First submitted 2018-07-13; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: pulmonary microbiota; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- exacerbating COPD patients needing ICU admission: sputum collection
  Interventions: Biological: Sputum collection

INTERVENTIONS:
Biological: Sputum collection — Analysis of Sputum collection

SUMMARY:
This study aims to investigate the correlation between pulmonary microbiota dynamics (including bacteria, fungi and viruses) and COPD exacerbation for COPD patients admitted to ICU

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a frequent cause of ICU admission. COPD exacerbations are a leading cause of lung function worsening and of morbimortality. Hospitalizations due to COPD exacerbations are highly expensive for health insurance system. Bacterial pulmonary microbiota has been shown to be correlated to the severity of COPD and to exacerbations. Nevertheless fungi and viruses which are full actors of pulmonary microbiota have not yet been investigated.

Our primary outcome will be the assessment of alpha and beta diversity dynamics of the whole pulmonary microbiota (bacteria, fungi and viruses) between COPD exacerbation and steady state.

This study will prospectively include 24 patients at ICU admission for COPD exacerbation with sputum sampling. Steady-state as defined during a 2 months-later visit will be studied with another sputum collection.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 admitted in ICU
* Admitted for COPD exacerbation defined by sustained (> 2 days) worsening of respiratory symptoms considering Anthonisen's criteria with life-threatening condition.
* Needing mechanical ventilation (noninvasive ventilation or oro-tracheal intubation)
* COPD condition will be presumed according to patient's respiratory history or previous lung function testing
* Able to consent or with the patient's family consent
* Affiliated to a social insurance scheme

No inclusion Criteria:

* COPD patient admitted for another cause than respiratory failure
* person under tutorship or curatorship
* living further than 100 kilometers away from the ICU
* expected survival inferior to 1 week

Exclusion Criteria

- Lung function testing not consistent with COPD at steady-state visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient above 18 admitted in ICU, admitted for COPD exacerbation defined by sustained (> 2 days) worsening of respiratory symptoms considering Anthonisen's criteria with life-threatening condition.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of differents types of cyto-bacteriological of sputum in Bacteriology | Day 0
  After extraction of the DNA and sequencing, the obtained sequences allow a taxonomic assignment of the microorganisms. The number of different taxonomic groups and the number of sequences within each taxonomic group to evaluate the α diversity through the coefficient developed by Shannon and the β diversity
Number of differents types of Cyto-bacteriological of sputum in Mycology | Day 0
  After extraction of the DNA and sequencing, the obtained sequences allow a taxonomic assignment of the microorganisms. The number of different taxonomic groups and the number of sequences within each taxonomic group to evaluate the α diversity through the coefficient developed by Shannon and the β diversity.
Number of differents types of Cyto-bacteriological of sputum in Virology | Day 0
  After extraction of the RNA and sequencing, the obtained sequences allow a taxonomic assignment of the microorganisms. The number of different taxonomic groups and the number of sequences within each taxonomic group to evaluate the α diversity and the β diversity.
Number of differents types of Cyto-bacteriological of sputum in Bacteriology | Day 60
  After extraction of the DNA and sequencing, the obtained sequences allow a taxonomic assignment of the microorganisms. The number of different taxonomic groups and the number of sequences within each taxonomic group to evaluate the α diversity through the coefficient developed by Shannon and the β diversity
Number of differents types of Cyto-bacteriological of sputum in Mycology | Day 60
  After extraction of the DNA and sequencing, the obtained sequences allow a taxonomic assignment of the microorganisms. The number of different taxonomic groups and the number of sequences within each taxonomic group to evaluate the α diversity through the coefficient developed by Shannon.
Number of differents types of Cyto-bacteriological of sputum in Virology | Day 60
  After extraction of the RNA and sequencing, the obtained sequences allow a taxonomic assignment of the microorganisms. The number of different taxonomic groups and the number of sequences within each taxonomic group to evaluate the α diversity and the β diversity.

CONTACTS AND LOCATIONS:
Overall Officials: Didier GRUSON, MD/PhD, Principal Investigator — Hospital University, Bordeaux
Locations (1):
- University Hospital, Bordeaux, Bordeaux, France